CLINICAL TRIAL: NCT06489951
Title: Efficacy and Mechanism of High-Dose Vitamin D Supplementation in Pediatric OAB-Dry: A Randomized Clinical Trial Integrating Urinary Myelin Basic Protein as a Theranostic Biomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xing Liu (Other)
Collaborators: Beijing Children's Hospital (Other); Shanghai Children's Hospital (Other); Children's Hospital of Soochow University (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xing Liu, Professor, Doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202453
Record Dates: First submitted 2024-06-24; First posted 2024-07-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder; Pediatric Disorder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Vitamin D

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Behavioral Therapy Combined with Solifenacin Drug Treatment (Experimental): Solinasine succinate 5mg once daily with a maximum dose of 10mg/day. Standard Behavioral Therapy
  Interventions: Drug: Solifenacin; Behavioral: Standard behavioral therapy
- Standard behavioral therapy combined with short-term high dose exogenous vitamin D supplementation (Experimental): Oral vitamin D drops, 2400iu/d, continued for 6 weeks after follow-up. Standard Behavioral Therapy
  Interventions: Dietary Supplement: vitamin D; Behavioral: Standard behavioral therapy

INTERVENTIONS:
Drug: Solifenacin — The outpatient physician prescribed Solinaxine (up to 0.5mg daily) to the participant orally
  Arms: Standard Behavioral Therapy Combined with Solifenacin Drug Treatment
Dietary Supplement: vitamin D — The outpatient physician prescribed vitamin d drops (2400iu daily) for the participants, which were taken orally by the participants
  Arms: Standard behavioral therapy combined with short-term high dose exogenous vitamin D supplementation
Behavioral: Standard behavioral therapy — Participants will receive an initial behavioral therapy session at enrollment and a second behavioral therapy session six weeks later. Education including information about dry OAB, lifestyle adjustments, bladder and pelvic floor training, bowel management, and how to use a bladder diary to record urination

SUMMARY:
The aim of this study is to give children with dry OAB: (1) Standard behavioral therapy combined with classical anticholinergic drugs (Solinaxine), or (2) standard behavioral therapy combined with short-term high-dose exogenous vitamin D supplementation are used to compare the outcomes of lower urinary tract symptoms in children with dry OAB during follow-up. To provide more robust supporting evidence for the broader promotion of short-term high-dose exogenous vitamin D supplements in combination with standard behavioral therapy as an effective treatment for dry OAB treatment in children.

ELIGIBILITY:
Inclusion Criteria:

1. Children older than 5 years who were admitted to the Department of Urology, Children's Hospital Affiliated to Chongqing Medical University and diagnosed with dry OAB.
2. The results of our laboratory indicated that the serum vitamin D level was lower than 35ng/mL.
3. The child (guardian) has been informed of the nature of the study, understands the provisions in the protocol, is able to guarantee compliance, and signs the informed consent.

Exclusion Criteria:

1. Patients with other urinary system malformations or serious diseases (such as hypospadias, cryptorchidism, posterior urethral valvular disease, vesicoureteral reflux, neurogenic bladder, urinary system tumors, urinary calculi, bladder and urethral injuries, etc.);
2. complicated with neurological diseases (such as epilepsy, spinal cord injury, spinal cord dysplasia, tethered cord syndrome, multiple sclerosis, autism spectrum disorder, etc.);
3. Patients with severe heart disease, abnormal liver and kidney function, lung disease, bone malformation, severe digestive tract disease, and genetic metabolic disease;
4. History of gastrointestinal surgery and urinary system surgery;
5. Dry stool, long-term constipation;
6. are taking anticonvulsant and antiepileptic drugs, hormones, antituberculosis drugs;
7. Previous history of hypercalcemia, hyperphosphatemia with renal rickets;
8. History of unexplained hematuria and urinary tract infection in the past 1 year;
9. Have a history of allergy or allergic reaction to vitamin D preparations;
10. Participating in another clinical study at the time of visit or during the follow-up of another clinical study;
11. Those who did not want to participate in the study or had poor follow-up compliance

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Change in daily urination frequency | week 1, week6，week 12
  To explore whether standard behavioral therapy combined with short-term high dose vitamin D (2400IU daily) is superior to standard behavioral therapy combined with anticholinergic drugs (Solinaxine) in improving the daily frequency of urination in children with dry OAB.

SECONDARY OUTCOMES:
Change in the mean urgency score | week 1, week6，week 12
  To explore whether standard behavioral therapy combined with short-term high dose exogenous vitamin D supplementation (2400IU daily) is superior to standard behavioral therapy combined with anticholinergic drugs (Solinaxine) in improving mean urinal urgency scores in children with dry OAB.
Change quality of life score | week 1, week6，week 12
  Quality of life scores are assessed on a scale of 0 to 3, where 0 indicates no impact on family, social or academic life; A score of 1 represents occasional effects; A score of 2 is a significant impact. A score of 3 indicates a serious impact on family, social or school life

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No